CLINICAL TRIAL: NCT00514332
Title: Etude Prospective Multicentrique randomisée Comparant Deux stratégies thérapeutiques Pour Les Cancers Coliques en Occlusion : stratégie Chirurgicale Exclusive Versus stratégie thérapeutique Avec Stent Colique Initial
Brief Title: Comparison Between Colorectal Stents and Primary Surgery in Obstructive Colonic Cancer. A Randomized, Controlled Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrolling participants stopped
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Toulouse (Other); University Hospital, Grenoble (Other); Rennes University Hospital (Other); University Hospital, Lille (Other); University Hospital, Angers (Other Government); University Hospital, Bordeaux (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF7683
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Colorectal Obstruction; Left Colonic Adenocarcinoma
Keywords: colorectal stents; colonic obstruction; colonic adenocarcinoma; colorectal surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): primary surgery group
  Interventions: Procedure: stent

INTERVENTIONS:
Procedure: stent — stent placement for colorectal cancer obstruction
  Other Names: self-expending metallic stents

SUMMARY:
To evaluate wether colorectal stenting carry a significant clinical advantage

DETAILED DESCRIPTION:
Randomized controlled comparison between stents and primary surgery in obstructive left colonic obstructive carcinoma outside palliative situations.

ELIGIBILITY:
Inclusion Criteria:

* obstructive stenosis due to left colorectal cancer

Exclusion Criteria:

* previous colorectal cancer
* other colorectal location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
number of stoma in each group | within the first 6 month(plus or minus 1 month) after surgery

SECONDARY OUTCOMES:
mortality in each group | within the first 6 month (plus or minus 1 month) after surgery
complications | within the first 6 month (plus or minus 1 month) after surgery
number of procedures | within the first 6 month (plus or minus 1 month) after surgery
length of stay | within the first 6 month (plus or minus 1 month) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand L MILLAT, MD-PhD, Principal Investigator — University Hospital, Montpellier

REFERENCES:
- [Derived] Pirlet IA, Slim K, Kwiatkowski F, Michot F, Millat BL. Emergency preoperative stenting versus surgery for acute left-sided malignant colonic obstruction: a multicenter randomized controlled trial. Surg Endosc. 2011 Jun;25(6):1814-21. doi: 10.1007/s00464-010-1471-6. Epub 2010 Dec 18. PMID 21170659